CLINICAL TRIAL: NCT07399795
Title: Citalopram Dose and the Risk of Serious Adverse Events in Older Adults With Low Kidney Function: A Population-Based Cohort Study Research Protocol
Brief Title: Citalopram and the Risk of Serious Adverse Events
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 2025 0906 615 000_2; ICES # 2025 0906 615 000_2 (Other: ICES)
Record Dates: First submitted 2026-01-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease (CKD); Elderly; Outpatient
Keywords: Chronic Kidney Disease; High-throughput computing; Drug Adverse Events; Selective Serotonin Reuptake Inhibitors; Citalopram; Elderly; Geriatrics; Drug Safety
MeSH Terms: conditions — Renal Insufficiency, Chronic; Drug-Related Side Effects and Adverse Reactions | interventions — Citalopram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low dose of Citalopram (10 mg/day): Residents of Ontario (and possibly Alberta), aged 66 years or older with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for Citalopram (low-dose 10 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to January 1, 2025, with a day supply of ≥7 days. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, and each patient will enter the cohort only once.
  Interventions: Drug: Citalopram 10 MG
- High dose of Citalopram (20 mg/day): Residents of Ontario (and possibly Alberta), aged 66 years or older with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for Citalopram (high-dose: 20 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to January 1, 2025, with a day supply of ≥7 days. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, and each patient will enter the cohort only once.
  Interventions: Drug: Citalopram 20 MG

INTERVENTIONS:
Drug: Citalopram 10 MG — The primary exposure of interest will be oral Citalopram at a dose of 10 or 20 mg/day.
  Groups: Low dose of Citalopram (10 mg/day)
Drug: Citalopram 20 MG — The primary exposure of interest will be oral Citalopram at a dose of 10 or 20 mg/day.
  Groups: High dose of Citalopram (20 mg/day)

SUMMARY:
This population-based cohort study aims to evaluate the safety of initiating a new outpatient prescription of citalopram at 20 mg/day (higher dose) compared to 10 mg/day (lower dose) in adults aged 65 years and older with reduced kidney function. The primary research question is whether initiating a higher dose of citalopram (20 mg/day) versus a lower dose (10 mg/day) in older adults with low kidney function (defined as an estimated glomerular filtration rate [eGFR] less than 45 mL/min per 1.73 m2, without dialysis or a history of kidney transplantation) is associated with an increased 30-day risk of a composite outcome comprising all-cause hospitalization, all-cause emergency department visits, or all-cause mortality.

DETAILED DESCRIPTION:
Many older adults experience mental health disorders, including depression and anxiety, in conjunction with reduced kidney function. Citalopram, a selective serotonin reuptake inhibitor, is frequently prescribed to this population for the treatment of depression and anxiety. However, both aging and impaired kidney function can result in elevated plasma concentrations of citalopram, increasing the risk of adverse events. Prescribing references, product monographs, and other standard sources provide inconsistent recommendations regarding initial dose adjustments for patients with low kidney function. This inconsistency may contribute to variable dosing practices in clinical settings, where many older adults with reduced kidney function are started on citalopram at a dose of 20 mg per day. Compared to a lower dose of 10 mg per day, this higher dose may be associated with increased rates of falls, fractures, gastrointestinal bleeding, arrhythmias, hospitalization, and mortality. Despite these potential risks, real-world evaluations remain limited. Recent analyses using a high-throughput approach with Ontario healthcare databases identified an increased risk of adverse outcomes in patients with advanced chronic kidney disease (CKD), defined as an estimated glomerular filtration rate (eGFR) less than 45 mL/min/1.73 m² without a history of dialysis or kidney transplant, who were newly prescribed citalopram compared to a cohort of non-users. To further investigate and validate these preliminary findings, a population-based retrospective cohort study is planned among older adults in Ontario, Canada. This study will assess the 30-day risk of serious adverse events following initiation of high versus low doses of citalopram in older adults with reduced kidney function, with the goal of informing safer prescribing practices.

Methods: This population-based retrospective cohort study will include older adults (aged 66 years or older) with an estimated glomerular filtration rate (eGFR) less than 45 mL/min/1.73 m2, who are not receiving dialysis and have no history of kidney transplantation. Participants will be identified from Ontario, and potentially Alberta, who have been dispensed a new outpatient prescription for oral citalopram (10 or 20 mg per day) with a minimum day supply of seven days. In Ontario, participant accrual will occur from January 1, 2008, to January 1, 2025. Based on the prescribed daily dose, individuals will be categorized into low-dose (10 mg/day) and high-dose (20 mg/day) groups. Propensity score weighting will be applied to balance baseline characteristics between groups. The primary outcome will be a 30-day composite of all-cause hospitalization, emergency department visit, or mortality. Objectives: The study will assess whether initiation of high-dose (20 mg/day) versus low-dose (10 mg/day) citalopram is associated with a higher 30-day risk of the composite outcome among older adults with reduced kidney function. Additionally, the study will evaluate whether baseline eGFR category modifies the risk of the 30-day composite outcome among patients initiating higher versus lower doses of citalopram in the outpatient setting. The cohort will be expanded to include all levels of baseline eGFR, and eGFR will be categorized as ≥60, 45-59, and <45 mL/min per 1.73 m².

Study Design and Setting: Data Sources: This study will use a population-based retrospective cohort design with linked administrative health data from Ontario, Canada. If the Ontario cohort does not provide sufficient sample size, Alberta health administrative data will be included using the same methodology. Ontario data will be sourced from ICES (ices.on.ca), which securely manages individual-level data for all Ontario residents covered by the province's single-payer healthcare system. Data use is authorized under section 45 of Ontario's Personal Health Information Protection Act, which does not require research ethics board review. The study will draw on several Ontario health databases: the Ontario Drug Benefit (ODB) for prescriptions, the Registered Persons Database (RPDB) for demographics and vital status, the Canadian Institute for Health Information Discharge Abstract Database (CIHI-DAD) and National Ambulatory Care Reporting System (NACRS) for hospitalizations and emergency visits, the Ontario Health Insurance Plan (OHIP) Database for physician billing, and the Ontario Laboratories Information System (OLIS) for laboratory data, including serum creatinine to estimate kidney function. If Alberta data are used, they will be accessed through the Alberta Kidney Disease Network (AKDN), with data available up to approximately 2021. The study protocol, including the description, design, and statistical analysis plan, will be publicly registered before outcome analyses. Results will be reported according to RECORD guidelines.

Study Population: All older adults (≥66 years) with an eGFR less than 45 mL/min per 1.73 m2, who are not receiving dialysis and have no history of kidney transplantation, and who received a new outpatient prescription for oral citalopram at an initial dose of 10 or 20 mg/day with a day supply of at least 7 days between 2008 and 2024, will be included. The dispensing date of the prescription will be defined as the index date. Only the first eligible prescription per individual will be included to ensure unique cohort entry. Each individual will enter the cohort only once. Patients will be classified as either "high-dose" or "low-dose" citalopram users.

Baseline Characteristics: Baseline variables will be obtained from health records, census files, hospital records, laboratory data, and physician claims. These variables will include demographic characteristics such as age, sex, rurality, and neighborhood income quintile, as well as comorbidities and medication use. Baseline comorbidities and healthcare utilization will be assessed using 5-year and 1-year look-back periods from the index date, respectively. Baseline medication use will be evaluated within 120 days prior to the index date. Eligible patients must have an outpatient serum creatinine measurement within 365 days prior to cohort entry to enable estimation of eGFR using the 2021 CKD-EPI equation. Patients with end-stage kidney disease, defined as those on dialysis or who have received a kidney transplant, will be excluded.

Outcomes: The primary outcome is the 30-day composite of all-cause hospitalization, emergency department visit, or mortality. Only the first hospitalization or emergency department visit within 30 days is counted. The components of the composite outcome are accurately coded in ICES data. The observation window begins on the prescription fill date and continues for 30 days. Loss to follow-up is expected to be less than 0.3%, as the observation period is under 90 days and annual provincial emigration in this age group is below 0.5%. Participant observation will be censored at the first occurrence of the outcome of interest, death (if not the outcome of interest), or 30 days after the index date, whichever occurs first.

Secondary outcomes will include the following: 1) Each component of the primary composite outcome, specifically 30-day all-cause hospitalization, all-cause emergency department visit, and all-cause mortality, analyzed separately. 2) A 30-day composite outcome of hospital admission or emergency department visit with delirium or encephalopathy (including disorientation, transient alteration of awareness, or other cognitive symptoms), or a hospital encounter involving an urgent computed tomography scan of the head. 3) A 30-day composite outcome of hospital admission or emergency department visit with fracture (hip, femur, humerus, wrist/forearm, pelvis, or spine), falls, hypotension, or syncope. 4) A 30-day hospital admission or emergency department visit with a composite outcome of atrial fibrillation/flutter, ventricular arrhythmia, or other arrhythmias (including pacemaker insertion, palpitations, unspecified tachycardia, atrioventricular block, supraventricular tachycardia, other conduction disorders, or implantable cardiac defibrillator).

Statistical analysis plan: Categorical variables will be reported as frequencies and proportions. Continuous variables will be presented as means with standard deviations (SD) or medians with interquartile ranges (IQR), as appropriate. Baseline characteristics will be compared between the high-dose (20 mg/day) and low-dose (10 mg/day) groups using standardized mean differences (SMDs). An absolute SMD greater than 10% will indicate a meaningful imbalance.

Balancing comparator group: Inverse probability of treatment weighting (IPTW) based on the propensity score will be used to balance baseline characteristics between the high-dose (20 mg/day) and low-dose (10 mg/day) groups, including all known predictors of citalopram use. Propensity scores will be estimated using a multivariable logistic regression model incorporating all baseline characteristics. The average treatment effect in the treated (ATT) weights will be applied, assigning patients in the low-dose group weights calculated as (propensity score / [1 - propensity score]), while patients in the high-dose group will receive a weight of 1. This approach will generate a weighted pseudo-sample of low-dose citalopram (10 mg/day) patients with a distribution of measured baseline characteristics similar to that of the high-dose citalopram (20 mg/day) group. Baseline characteristics will be compared between groups using standardized differences in both unweighted and weighted samples. Regression analysis: To assess the primary composite outcome of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality, a modified Poisson regression will be used to estimate the risk ratio (95% CI), and binomial regression will be used to estimate the risk difference (95% CI) in the weighted cohort, with the low-dose citalopram (10 mg/day) group as the referent. Secondary analyses: All secondary outcomes will be tested independently without adjustment for multiple comparisons. Each test will be conducted and reported separately. Consistent with best practices, the primary outcome will be presented with its P-value, and all secondary outcomes will be reported as point estimates with 95% confidence intervals.

Additional analyses: Five supplementary analyses are planned. 1. Effect measure modification (EMM): The cohort will be expanded to include all estimated glomerular filtration rate (eGFR) levels, categorized into three groups: eGFR ≥60, 45-<60, and <45 mL/min/1.73 m². Baseline characteristics between high-dose (20 mg/day) and low-dose (10 mg/day) citalopram groups will be assessed using standardized differences for all renal function categories combined and within each eGFR category. To balance baseline characteristics between high-dose and low-dose citalopram groups, the inverse probability of treatment weighting (IPTW) method, based on propensity scores, will be applied for all eGFR categories combined and within each category. EMM will be evaluated on both additive and multiplicative scales. For additive interaction, binomial regression with an identity link will be used to estimate risk differences, including an interaction term between dose groups and eGFR strata. For multiplicative interaction, modified Poisson regression will estimate risk ratios, including an interaction term between dose groups and eGFR strata. The estimated risk difference and risk ratio will be reported as point estimates with their 95% CI in the subgroups. 2. A high-throughput computing analysis involving over 700 population-based, new-user cohort studies, each comparing 74 acute (30-day) outcomes across kidney function strata (PMID: 38186562), suggested that citalopram use versus no use is associated with harm in patients with low kidney function. This analysis used Ontario data from January 1, 2008 to March 1, 2020. A subgroup analysis will restrict the cohort to periods before March 1, 2020 (overlapping with the high-throughput computing period) and after March 1, 2020 (no overlap). 3. Hazard ratios for all outcomes within 30 days will be computed to illustrate the effect of the intervention over time. Hazard ratios are expected to be similar to risk ratios. 4. E-value analyses will be performed to determine the minimum association strength an unmeasured confounder would require with both the prescription drug and the outcome to eliminate the observed association. 5. The risk of the primary outcome will be compared between new users of 20 mg/day of citalopram and older adults with no citalopram use (non-users). The same comparison will be conducted for new users of 10 mg/day of citalopram versus non-users. The same baseline characteristics and statistical analysis methods as in the primary analysis will be employed.

*This approach will be implemented only if analysis of Alberta data proceeds.* Due to privacy regulations in Canada, individual-level patient data from different provinces cannot be linked. Instead, results from Ontario and Alberta will be combined using a privacy-preserving method to ensure data privacy and regulatory compliance. The proposed approach involves a single transfer of summary-level outputs from each province to the research team and will be adapted from the techniques described by Shu et al. 2025.

ELIGIBILITY:
Inclusion Criteria:

* Older adult aged 66 years or greater with low kidney function (an eGFR <45 mL/min per 1.73 m2 ) who have filled a new oral prescription for Citalopram at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program with a dose of 10 or 20 mg/day and a day supply of ≥7 days from January 1, 2008, to January 1, 2025 for Ontario (if needed, dates in Alberta to be finalized based on data availability). The investigators will exclude individuals undergoing dialysis or those who have received a kidney transplant. The age criterion is set to guarantee that individuals in this population had at least one year of prior universal outpatient prescription drug coverage. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once.

Exclusion Criteria:

1. Individuals with missing administrative database number, missing or invalid age (<0 or >105 years), missing or invalid sex, death on or before the index date, non-Ontario resident (for Ontario data).
2. Individuals less than 66 years of age on the index date.
3. Those with evidence of any study drug prescription 180 days before the index date (to restrict to new users only).
4. Individuals with other Selective Serotonin Reuptake Inhibitors (Escitalopram, Fluoxetine, Fluvoxamine, Paroxetine, Sertraline) prescription in the previous 180 days before the index date or on the index date.
5. Individuals with more than one study drug prescription on the index date, as this complicates the ability to ascertain the prescribed dose accurately.
6. Individuals with end-stage renal disease, chronic dialysis, or a kidney transplant prior to the index date.
7. Evidence with hospital discharge or emergency department visit in the two days prior to or on the index date to ensure a new outpatient prescription.
8. Individuals with no serum creatinine lab value in the 0-365 days prior to the index date.
9. Individuals with unstable baseline kidney function:• If the most recent serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] (refer to this as test date 1), and there is not at least one 'outpatient' serum creatinine in the year before test date 1, OR• If the most recent prior serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] (refer to this as test date 1), and while there is at least 'outpatient' serum creatinine test in the year before (test date 1), the most recent outpatient test prior to (test date 1) differs by an eGFR 10 mL/min/1.73 m2 or more from the value on (test date 1). In Ontario, it has been shown that an outpatient serum creatinine measurement in the province, conducted on a single occasion, usually represents a stable value.
10. Individuals receiving palliative care in the year prior to the index date, as in this setting dosing is less relevant; rather, the focus is comfort care. The investigators will restrict to the first prescription in individuals with more than one eligible prescription. Date of this prescription will be the index date (the date from which the outcomes start being assessed).

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population includes adults aged 66 years or older with reduced kidney function (eGFR less than 45 mL/min per 1.73 m2, excluding individuals receiving dialysis or with a history of kidney transplantation) who initiated a new outpatient prescription for Citalopram at a dose of 10 or 20 mg per day, with a minimum day supply of seven days, between 2008 and 2024 in Ontario. The accrual period for Alberta will be established based on data availability, if required.
Sampling Method: Non-Probability Sample
Enrollment: 7110 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01 (Actual)

PRIMARY OUTCOMES:
A composite outcome of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality. | From cohort entry (Day 0) through 30 days post-entry or until first event (hospitalization, ED visit, or death), whichever occurs first.
  All-cause hospitalization, all-cause emergency department visits, and all-cause mortality will be combined into a composite measure. Only the first hospitalization or first emergency department visit occurring after the cohort entry date will be considered.

SECONDARY OUTCOMES:
All-cause hospitalization | From cohort entry (Day 0) through 30 days post-entry or until first event (hospitalization, ED visit, or death), whichever occurs first.
  One of the components of the primary composite outcome, all-cause hospitalization, individually presented as a secondary outcome. Only the first hospitalization after the cohort entry date will be considered.
All-cause emergency department visit | From cohort entry (Day 0) through 30 days post-entry or until first event (hospitalization, ED visit, or death), whichever occurs first.
  One of the components of the primary composite outcome, all-cause emergency department visit, individually presented as a secondary outcome. Only the first emergency department visit after the cohort entry date will be considered.
All-cause mortality | From cohort entry (Day 0) through 30 days post-entry or until first event (hospitalization, ED visit, or death), whichever occurs first.
  One of the components of the primary composite outcome, all-cause mortality, individually presented as a secondary outcome.

OTHER OUTCOMES:
30-day hospital encounter with composite outcome of Atrial Fibrillation/flutter or ventricular arrhythmia or other arrhythmia | Through 30 days after cohort entry
  30-day hospital encounter (hospital admission or emergency visit) composite of atrial fibrillation/flutter or ventricular arrhythmia, or other arrhythmia (including pacemaker insertion, palpitations, tachycardia unspecified, atrioventricular block, supraventricular tachycardia, other conduction disorders, implantable cardiac defibrillator)
30-day composite outcome of a hospital encounter with delirium, encephalopathy, or hospital encounter with receipt of an urgent computed tomography scan of the head | Through 30 days after cohort entry
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with delirium or encephalopathy (disorientation, transient alteration of awareness, other and unspecified symptoms and signs involving cognitive function) or hospital admission with receipt of an urgent computed tomography scan of the head.
30-day composite outcome of a hospital encounter with fracture, falls, hypotension, or syncope | Through 30 days after cohort entry
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with fracture, falls, hypotension, or syncope.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Garg, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute
Locations (1):
- London Health Sciences Centre Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The dataset in Ontario from this study is held securely in coded form at ICES. While legal data sharing agreements between ICES and data providers (e.g., healthcare organizations and government) prohibit ICES from making the dataset publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at www.ices.on.ca/DAS (email: das@ices.on.ca). The full dataset creation plan and underlying analytic code may be available from the authors for a certain period of time after the study is completed upon request, understanding that the computer programs may rely upon coding templates or macros that are unique to ICES and are therefore either inaccessible or may require modification.

REFERENCES:
- [Background] Abdullah SS, Rostamzadeh N, Muanda FT, McArthur E, Weir MA, Sontrop JM, Kim RB, Kamran S, Garg AX. High-Throughput Computing to Automate Population-Based Studies to Detect the 30-Day Risk of Adverse Outcomes After New Outpatient Medication Use in Older Adults with Chronic Kidney Disease: A Clinical Research Protocol. Can J Kidney Health Dis. 2024 Jan 6;11:20543581231221891. doi: 10.1177/20543581231221891. eCollection 2024. PMID 38186562